CLINICAL TRIAL: NCT03341598
Title: Comparison of Different Surgical Approaches for Root Coverage of Teeth Presenting With Gingival Recession Associated With Non-carious Cervical Lesion Partially Restored With Composite Resin. Randomized Controlled Clinical Trial
Brief Title: Two Surgical Approaches for Root Coverage of Teeth Presenting Gingival Recession and Non-carious Cervical Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEPJMF 8
Record Dates: First submitted 2017-05-11; First posted 2017-11-14 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Filtek Supreme

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF+R (Active Comparator): First of all, a sterile rubber dam will be placed to isolate the operative field and the non-carious cervical lesion restoration was performed with a nanocomposite resin (Filtek Supreme - 3M- St. Paul, Minnesota, USA), following the manufacturer's instructions. CAF treatment will be performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision will be made to unite the releasing incisions and the flap will be raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Sling sutures will be placed to stabilize the flap in a coronal position 2 mm above the cementoenamel junction (CEJ), followed by interrupted sutures to close the releasing incisions.
  Interventions: Procedure: CAF; Procedure: R
- CAF+R+MC (Experimental): First of all, a sterile rubber dam will be placed to isolate the operative field and the non-carious cervical lesion restoration was performed with a nanocomposite resin (Filtek Supreme - 3M - St. Paul, Minnesota, USA), following the manufacturer's instructions. CAF treatment will be performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision will be made to unite the releasing incisions and the flap will be raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Additionally, this group will receive the xenogenous collagen matrix graft (Geistlich) on the recessed area before the sutures. Then, the flap will be coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: CAF; Procedure: R; Procedure: MC

INTERVENTIONS:
Procedure: CAF — Periodontal surgical technique to treat gingival recessions.
  Other Names: Periodontal plastic surgery
Procedure: R — Restorative procedure to treat tooth structure loss.
  Other Names: Composite resin restoration (Filtek Supreme - 3M)
Procedure: MC — Xenogenous graft placed in the surgical site.
  Other Names: Xenogenous collagen matrix
  Arms: CAF+R+MC

SUMMARY:
The aim of the present study is to compare the use of the xenogeneic graft (MC) plus coronary advanced flap (CAF) and the coronary advanced flap alone, both associated with the partial restoration of composite resin in the treatment of gingival recessions associated with non-carious cervical lesion.

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial. The population evaluated in the study was selected at Institute of Science and Technology (ICT), São José dos Campos, College of Dentistry.

Sixty patients presenting gingival recession will be divided in 2 groups:

* Group 1 - Test: 30 gingival recessions associated with non-carious cervical lesions that will receive partial composite resin restoration and periodontal surgery for root coverage through a xenogenic collagen matrix graft (CAF + MC + R)
* Group 2 - control: 30 gingival recessions associated with non-carious cervical lesions that will receive partial composite resin restoration and periodontal surgery for root coverage (CAF + R) without graft.

The surgeries, as well as all postoperative follow-up, were performed at the dental clinic of ICT. Two horizontal incisions were made at right angles to the adjacent interdental papillae, without interfering with the gingival margins of neighboring teeth. Two oblique vertical incisions were extended beyond the mucogingival junction, and a trapezoidal mucoperiosteal flap was raised up to the mucogingival junction. After this point, a split-thickness flap was extended apically, releasing the tension and favoring coronal positioning of the flap.The exposed root surface was gently scaled and planed until it became smooth in the connective tissue graft (CTG) group. For those allocated to CTG plus composite resin (CR) group, a sterile rubber dam was placed to isolate the operative field and the non-carious cervical lesion restoration was performed with a nanocomposite resin (Filtek Supreme - 3M - St. Paul, Minnesota, USA), following the manufacturer's instructions. Afterward, the both groups received a thin and small connective tissue graft that was sutured over the root/restoration surface. Then, the flap was coronally positioned and sutured to completely cover the graft.

Clinical parameters were assessed at baseline and 3 and 6 months post-operatively.

Statistical Analysis The null hypothesis considered in the study was the absence of difference in the clinical parameters between the different groups. For data analysis, the statistical program was used (SigmaPlot). The demographic and clinical data were compared between the groups using Student's t-test. The data were first analyzed for homogeneity using the Shapiro-Wilk test, which indicated non-normal distribution. . Those presenting Shapiro-Wilk p values < 0.05 were analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Patients' esthetics and discomfort measures using a visual analog scale (VAS) were analyzed by T-tests. The frequency of sites that were scored as very good or excellent in each group by qualitative cosmetic evaluation (QCE) analysis, the frequency of complete root coverage, bleeding on probing (BOP), and the presence or absence of plaque at the site were compared using χ2 tests. Intergroup root esthetic scale (RES) comparisons were performed with a T-test. A significance level of 0.05 was adopted.

ELIGIBILITY:
Inclusion Criteria:

* presenting Miller class I or II gingival recession in the maxillary canines or premolars associated with non-carious cervical lesion;
* teeth included in the study should present pulp vitality;
* patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤ 20%;
* patients older than 18 years old;
* probing depth ˂ 3 mm in the included teeth;
* patients who agreed to participate and signed an informed consent form

Exclusion Criteria:

* patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure
* patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure
* smokers or pregnant women
* patients who underwent periodontal surgery in the area of interest;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Recession reduction | 1 year
  Recession reduction from baseline measured in millimetres

SECONDARY OUTCOMES:
Root coverage esthetic score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP
Locations (1):
- São Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zucchelli G, Gori G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Non-carious cervical lesions associated with gingival recessions: a decision-making process. J Periodontol. 2011 Dec;82(12):1713-24. doi: 10.1902/jop.2011.110080. Epub 2011 May 4. PMID 21542735
- [Background] Santamaria MP, Fernandes-Dias SB, Araujo CF, Lucas da Silva Neves F, Mathias IF, Rebelato Bechara Andere NM, Neves Jardini MA. 2-Year Assessment of Tissue Biostimulation With Low-Level Laser on the Outcomes of Connective Tissue Graft in the Treatment of Single Gingival Recession: A Randomized Clinical Trial. J Periodontol. 2017 Apr;88(4):320-328. doi: 10.1902/jop.2016.160391. Epub 2016 Nov 11. PMID 27834120
- [Derived] Mathias-Santamaria IF, Silveira CA, Rossato A, Sampaio de Melo MA, Bresciani E, Santamaria MP. Single gingival recession associated with non-carious cervical lesion treated by partial restoration and coronally advanced flap with or without xenogenous collagen matrix: A randomized clinical trial evaluating the coverage procedures and restorative protocol. J Periodontol. 2022 Apr;93(4):504-514. doi: 10.1002/JPER.21-0358. Epub 2021 Aug 21. PMID 34310715